CLINICAL TRIAL: NCT01374217
Title: Administration of an Oral PDE5 Inhibitor, Tadalafil in Conjunction With Lenalidomide and Dexamethasone in Patients With Multiple Myeloma
Brief Title: Administration of Tadalafil in Conjunction With Lenalidomide and Dexamethasone in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: early stopping rule
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1167; NA_00049238 (Other: JHMI IRB)
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Tadalafil; Lenalidomide; Dexamethasone; Calcium Dobesilate; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tadalafil (Experimental): Subject will take tadalafil in combination with with Lenalidomide and dexamethasone (Rd) or Clarithromycin/Lenalidomide/ dexamethasone (BiRd)
  Interventions: Drug: Tadalafil; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Clarithromycin

INTERVENTIONS:
Drug: Tadalafil — Tadalafil will be administered at a dose of 20 mg orally daily starting with day 1 of the first cycle. Each cycle will last for 28 days
  Other Names: Cialis
Drug: Lenalidomide — Lenalidomide will be administered as it was prior to study entry.
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone will be administered as it was prior to study entry.
  Other Names: Decadron
Drug: Clarithromycin — Clarithromycin will be administered as it was prior to study entry.
  Other Names: Biaxin

SUMMARY:
The primary objective of this study is to evaluate the anti-tumor efficacy of tadalafil in combination with Lenalidomide/dexamethasone (Rd) in multiple myeloma.

DETAILED DESCRIPTION:
This is an early phase study to evaluate the safety and efficacy of the combination of tadalafil with lenalidomide and dexamethasone (Rd) or BiRd. 19 patients on Rd or BiRd will be treated with tadalafil for a minimum of 6 months. The investigational drug will be discontinued if there is evidence of disease progression as defined by the International Uniform Response criteria [1]. For responding patients (patients who have a CR, VGPR, PR or SD), the therapy will be continued until progression or intolerable adverse effects. Blood and bone marrow will be collected for various studies as detailed in section 14.10. Clinical response will be monitored every month during the study.

ELIGIBILITY:
Inclusion Criteria:

* Progressive myeloma as defined by the International Uniform Criteria.
* Currently on Lenalidomide and dexamethasone for the treatment of myeloma
* Age > 18 years.
* Measurable paraprotein in serum or urine or detectable free light chains in the serum.
* ECOG performance status of 0 - 2.

Exclusion Criteria:

* Hypersensitivity to PDE5 inhibitors such as tadalafil, sildenafil or vardenafil.
* History of malignancy other than multiple myeloma in the last five years of, except adequately treated basal or squamous cell skin cancer.
* Participation in any clinical trial which involved an investigational drug or device four weeks prior.
* Infection requiring treatment with antibiotics, antifungal, or antiviral agents in the last seven days
* Any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
* History of significant hypotensive episode requiring hospitalization.
* Acute myocardial infarction within prior 3 months, uncontrolled angina
* Uncontrolled arrhythmia, or uncontrolled congestive heart failure
* History of any of the following cardiac conditions:

I. Angina requiring treatment with long-acting nitrates. II. Angina requiring treatment with short-acting nitrates within 90 days of planned tadalafil administration.

III. Unstable angina within 90 days of visit 1. IV. Positive cardiac stress test without documented evidence of subsequent, effective cardiac intervention.

- History of any of the following coronary conditions within 90 days of planned tadalafil administration:

i. Myocardial Infarction.

ii. Coronary artery bypass graft surgery.

iii. Percutaneous coronary intervention (for example, angioplasty or stent placement).

iv. Any evidence of heart disease (NYHA≥Class III) within 6 months of planned tadalafil administration.

* Current treatment with nitrates.
* Current systemic treatment with a potent cytochrome P450 3A4 (CYP3A4) inhibitors such as ketoconazole or ritonavir.
* Prior chronic immune suppressive state (AIDS, immunosuppressive therapy).
* History of hypotension and/or blindness or sudden decrease/loss of hearing during prior treatment with PDE-5 inhibitors.
* Prior history of non-arterial ischemic optic retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilanjan Ghosh, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was a screen failure.
Period: Overall Study
Arm/Group | Tadalafil
Started | 13
Completed | 0
Not Completed | 13
Not completed — Lack of Efficacy | 13

BASELINE CHARACTERISTICS:
Arm/Group | Tadalafil
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 5
Age, Continuous [Median (Full Range); unit: years] | 63 [52 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Percentage of participants who responded to the addition of tadalafil. Response is defined as a complete remission (CR), very good partial remission (VGPR), partial remission (PR), or stable disease (SD) by International Uniform Response criteria.
Time Frame: Up to 6 months
Population: One participant was not analyzed because he only received eight days of study drug prior to progression and removal from study. One participant was retrospectively ineligible and was therefore not analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Tadalafil
Number analyzed (Participants) | 11
Participants | 5

2. Secondary Outcome: Duration of Response
Description: Median length of response in months.
Time Frame: Up to 6 months
Population: This analysis only includes the 5 participants who had a clinical response.
Measure: Median (Full Range); unit: months
Arm/Group | Tadalafil
Number analyzed (Participants) | 5
months | 2.3 [1.6 to 5.3]

3. Secondary Outcome: Time to Progression
Description: Median time to progression of disease in days.
Time Frame: Up to 71 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tadalafil
Number analyzed (Participants) | 11
days | 48 [25 to 71]

4. Secondary Outcome: Quality of Life Scores
Description: Median change in symptom scores. Scale is the EORTC QLQ-C30. There are three domains: symptom scale (score range 7-14); past week (score range 21-82); and global health status (score range 2-14). Higher or increasing scores mean worse outcomes; lower or decreasing scores mean better outcomes.
Time Frame: 3 months (M3) and 6 months (M6)
Population: Two participants returned the Month 3 survey and seven participants returned the Month 6 survey (there is some overlap). The remaining participants cannot be analyzed as there is no follow-up data.
Measure: Median (Full Range); unit: change in score on a scale
Arm/Group | Tadalafil
Number analyzed (Participants) | 8
change in score on a scale
  Symptoms (M3): number analyzed (Participants) | 2
  Symptoms (M3) | 0 [0 to 0]
  Past week (M3): number analyzed (Participants) | 2
  Past week (M3) | 5 [-1 to 11]
  Global health status (M3): number analyzed (Participants) | 2
  Global health status (M3) | -1.5 [-3 to 0]
  Symptoms (M6): number analyzed (Participants) | 7
  Symptoms (M6) | 1 [-1 to 3]
  Past week (M6): number analyzed (Participants) | 7
  Past week (M6) | 6 [-4 to 9]
  Global health status (M6): number analyzed (Participants) | 7
  Global health status (M6) | -1 [-7 to 0]

5. Secondary Outcome: Effect of PDE5 Inhibition on Immune Function as Assessed by MDSC Quantification
Description: Percentage change in the amount of myeloid derived suppressor cells (MDSCs) in peripheral blood.
Time Frame: Up to 6 months
Population: Data was not collected to assess this outcome measure.
Arm/Group | Tadalafil
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 7 months
Description: Adverse events were collected monthly.
Arm/Group | Tadalafil
All-Cause Mortality (participants affected / at risk) | 6/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=13)
Anorexia (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurred vision (Nervous system disorders) | 1 (1)
Cold intolerance (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Dizziness (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Eye floaters (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 9 (11)
Fever (Infections and infestations) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
GI bleed (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (4)
High creatinine (Investigations) | 1 (1)
Hyperglycemia (Investigations) | 8 (14)
Hypoalbuminemia (Investigations) | 2 (3)
Hypocalcemia (Investigations) | 4 (9)
Hypokalemia (Investigations) | 2 (2)
Insomnia (Nervous system disorders) | 2 (2)
Lymphopenia (Investigations) | 7 (22)
Neutropenia (Investigations) | 10 (22)
Low carbon dioxide (Investigations) | 1 (1)
Anemia (Investigations) | 13 (33)
Thrombocytopenia (Investigations) | 9 (23)
Leukopenia (Investigations) | 11 (25)
Impaired memory (Nervous system disorders) | 2 (2)
Mucositis (Gastrointestinal disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Neuropathy (Nervous system disorders) | 6 (9)
Neutropenic fever (Infections and infestations) | 1 (1)
Night sweats (General disorders) | 2 (2)
Epistaxis (General disorders) | 1 (1)
Osteonecrosis of the jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - back (Musculoskeletal and connective tissue disorders) | 7 (12)
Pain - bone (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - hip (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - rib (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - throat (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Red eyes (Eye disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Hallucinations (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight gain (General disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Xerosis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No